CLINICAL TRIAL: NCT01074203
Title: A Pilot Study to Explore a Potential Role of Nitazoxanide (NTZ) in the Prevention of Recurrent Hepatitis C Virus (HCV) Infection After Orthotopic Liver Transplantation
Brief Title: A Pilot Study to Examine the Role of Nitazoxanide to Prevent Recurrence of Hepatitis C After Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: W Ray Kim, Mayo Clinic College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 08-006000
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Hepatitis C Recurrence
Keywords: nitazoxanide; liver transplantation; HCV recurrence
MeSH Terms: interventions — nitazoxanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitazoxanide arm (Experimental): All patients will receive nitazoxanide
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide — Drug administration: The drug will be available through the research pharmacy. Patients will receive 1000mg (2 tablets) oral NTZ or an equivalent dose of NTZ suspension 1500mg (75mL) according to the schedule below.
  Dose timing Dose Schedule Interval Dose Pre-transplant(on admission) 1000mg oral Once Total 1 dose Pre-transplant (delayed surgery >12 hours) 1000mg oral Every 12 hrs Variable Post operative dose 1000mg oral/ nasogastric tube Every 12 hrs Total 6 doses
  All attempts will be made to administer the tablet form of the medication, given the higher area under the curve that is achieved. If needed, the suspension formulation will be used. Since the suspension form has 70% bioavailability, the suspension dose administered will be 1.5 grams every 12 hours until the tablet form can be given.

SUMMARY:
Recurrence of Hepatitis C virus infection (HCV) is universal after orthotopic liver transplantation (LTx) and is associated with allograft failure, death and need for re-transplantation. Currently, there are no effective therapies to prevent HCV recurrence. Nitazoxanide (NTZ), an oral thiazolide anti-infectious agent, was safe, well tolerated and effective in achieving sustained viral response in patients with chronic HCV genotype 4. Its role in the prevention of HCV recurrence after liver transplantation has not been studied. The investigators propose to conduct an open label pilot study examining the role of NTZ in the prevention of HCV re-infection in eight patients undergoing LTx. First time transplant recipients for chronic HCV without history of renal failure or HIV/HBV co-infection, will receive NTZ immediately prior to LTx and for 3 days thereafter. The primary endpoint is the number of patients who remain HCV-RNA-negative at day 7 after LTx. If at least one patient remains negative, the study will be determined to be positive. Additionally, the investigators will examine the viral kinetics of HCV, tolerability and safety of NTZ.

DETAILED DESCRIPTION:
Recurrence of Hepatitis C virus infection (HCV) is universal after orthotopic liver transplantation (LTx) and is associated with allograft failure, death and need for re-transplantation. Currently, there are no effective therapies to prevent HCV recurrence. Nitazoxanide (NTZ), an oral thiazolide anti-infectious agent, was safe, well tolerated and effective in achieving sustained viral response in patients with chronic HCV genotype 4. Its role in the prevention of HCV recurrence after liver transplantation has not been studied. We propose to conduct an open label pilot study examining the role of NTZ in the prevention of HCV re-infection in eight patients undergoing LTx. First time transplant recipients for chronic HCV without history of renal failure or HIV/HBV co-infection, will receive NTZ immediately prior to LTx and for 3 days thereafter. The primary endpoint is the number of patients who remain HCV-RNA-negative at day 7 after LTx. If at least one patient remains negative, the study will be determined to be positive. Additionally, we will examine the viral kinetics of HCV, tolerability and safety of NTZ.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients age 18-75
* HCV infection identified by positive, quantifiable HCV RNA prior to transplant

Exclusion Criteria:

* Scheduled recipient of living donor transplantation
* History of chronic hepatitis B or HIV infection
* Transplantation for fulminant hepatic failure
* Estimated glomerular filtration rate <60ml/min
* Women who are pregnant or breast feeding and men or women that are sexually active but do not agree to use acceptable birth control

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
undetectable HCV RNA by real-time reverse transcription PCR on day 7 after transplantation. | at day 7
  undetectable HCV RNA by real-time reverse transcription PCR on day 7 after transplantation.

SECONDARY OUTCOMES:
Viral Kinetics | 4 months
  Viral Kinetics: The decline in HCV RNA will be calculated using the HCV RNA levels obtained during the study at the 12 time points.
Safety | 7 days
  Safety of NTZ: The safety and tolerability of NTZ will be monitored by evaluating vital signs, change in laboratory data from baseline, adverse events, UPIRSTOs, dose adjustments and incidence of early drug withdrawal. Tolerability will be defined as the number of patients discontinuing medications or having a dose modification due to an adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: W Ray Kim, MD, Principal Investigator — Mayo Clinic College of Medicine
Locations (1):
- Mayo Clinic College of Medicine, Rochester, Minnesota, United States